CLINICAL TRIAL: NCT01135771
Title: Performance Study Using the OptiScanner on Healthy Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: OptiScan Biomedical Corporation (Industry)
Responsible Party: Dr. Tim Heise, Profil Institut für Stoffwechselforschung GmbH
Masking: None | Purpose: Diagnostic
Other Study IDs: 1003106
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes
Keywords: glucose monitoring; diabetes; glucose monitoring in patients with diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: glucose and insulin IV to alter blood glucose

SUMMARY:
This study is designed to demonstrate the accuracy of the OptiScanner glucose measurement. The accuracy of the test device will be determined using plasma samples collected directly from Type 1 and Type 2 Diabetics using the OptiScanner. Blood samples will simultaneously be collected and measured on YSI 2300 STAT PLUS (YSI) made by YSI Incorporated. These results will be compared to the OptiScanner's glucose measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed an Informed Consent Form for this study approved by the Institutional Review Board (IRB)
2. Have a documented onset of diabetes ³ 1 year prior to this study
3. Have Type 1 or Type 2 diabetes according to the American Diabetes Association diagnostic criteria
4. Be currently treated with insulin (all regimens) for ³ 1 year and able (as judged by Investigator) and willing to undergo a hypoglycemic challenge and a hyperglycemic challenge; oral diabetes medication in combination with insulin is allowed
5. Be at least 18 but no more than 65 years of age
6. Be willing and able to comply with the requirements of the protocol
7. Be willing to refrain from participating in any other investigational study while enrolled in this study
8. For Female Subjects: Be post-menopausal, sterilized or not of child-bearing potential, or have a negative pregnancy test and have no intention of becoming pregnant between Visit 1 and Visit 2, and be using contraceptive devices or drugs (risk of pregnancy must be lower than 1%).

Exclusion Criteria:

1. Recurrent major hypoglycemia (as judged by the Investigator) or hypoglycemia requiring hospitalization within the last 12 months
2. Have a history of hypoglycemic seizure within the last year
3. Impaired hepatic function measured as AST/ALT ³ two and a half times the upper reference limit or total bilirubin two and a half times the upper reference limit based on analysis from the local laboratory, or at the Investigator's discretion
4. Impaired renal function measured as creatinine ³ 1.5 (females) mg/dL, ³ 1.7 (males) mg/dL based on analysis from the local laboratory, or at the Investigator's discretion
5. Haematocrit or electrolytes (sodium, potassium) outside of normal limits based on analysis from the local laboratory, or at the investigator's discretion.
6. Have Uric Acid > 10 mg/dL based on analysis from the local laboratory
7. HIV positive, or Hepatitis B or C positive (blood test required). A viral load test will be done at the local laboratory for subjects with a positive Hepatitis result.
8. New York Heart Association (NYHA) Class III or IV congestive heart failure
9. Have a history of angina requiring hospitalization or a myocardial infarction within the last 12 months
10. Evidence of intermittent or sustained ventricular or supra-ventricular arrhythmias such as ventricular tachycardia, atrial fibrillation, etc. Holter monitoring may be performed to exclude arrhythmias at the discretion of the investigator.
11. Uncontrolled treated/untreated hypertension (systolic blood pressure ³ 160 mmHg and/or diastolic blood pressure ³ 100 mmHg)
12. Have active diabetic proliferative retinopathy (undergoing treatment)
13. Have active significant recurring skin infections or adhesive allergies, at the Investigator's discretion
14. Have given more than 150 mL of blood within 8 weeks prior to enrollment in this study
15. Currently taking anticoagulants, e.g. Coumadin (warfarin), Marcumar (phenprocoumon). Patients with prolonged activated PTT will not be included in this study.
16. Have received any investigational product or been treated with an invasive device within the past 30 days
17. Mental incapacity, unwillingness or language barrier precluding adequate understanding or co-operation
18. Any chronic illness that, in the judgment of the Investigator, may hinder or confuse compliance with the protocol
19. Any condition (may include clinically significant screening laboratory assessments) which, in the judgement of the Investigator, may increase the risk to the subject or decrease the likelihood of achieving the objectives of the study
20. Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
demonstrate the accuracy of the OptiScanner in measuring blood glucose levels in otherwise healthy diabetic subjects when compared to blood glucose levels simultaneously measured on the YSI

SECONDARY OUTCOMES:
The secondary objective of the study is to demonstrate a blood glucose measurement range of 60 to 500 mg/dL at the hematocrit levels referenced as normal

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, Germany

REFERENCES:
- See also: Related Info — http://www.profil.com